CLINICAL TRIAL: NCT02873156
Title: A Randomized, Double-Blind, Placebo-Controlled, Multiple Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of E2027 in Healthy Subjects
Brief Title: A Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of E2027 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: E2027-A001-002
Record Dates: First submitted 2016-08-16; First posted 2016-08-19 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2017-11

CONDITIONS: Healthy Subjects
Keywords: E2027; Healthy participants; Pharmacokinetics; Pharmacodynamics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (2):
- E2027 (Experimental): Four sequential cohorts of healthy participants (≥50 years and ≤85 years old) will be treated with multiple ascending doses of E2027 up to the maximum tolerated dose (MTD). A total of 6 participants per cohort will be randomized to E2027.Proposed doses of E2027 are:
  * Part A Cohort 1: 50 mg (1 × 50 mg capsule)
  * Cohort 2: 100 mg (2 × 50 mg capsules)
  * Cohort 3: 200 mg (4 × 50 mg capsules)
  * Cohort 4: 400 mg (8 × 50 mg capsules)
  * Cohort 6: 25 mg (5 × 5 mg capsules) Part B
  * Cohort 5: 400 mg (8 × 50 mg capsule)
  Part C:
  • Cohort 7: 50 mg (1 × 50 mg capsules)
  Part D:
  * Cohort 8: 5 mg (1 × 5 mg capsules)
  * Cohort 9: 10 mg (2 × 5 mg capsules)
  Interventions: Drug: E2027
- Placebo (Placebo Comparator): Four sequential cohorts of healthy participants (≥50 years and ≤85 years old) will be treated with multiple ascending doses of E2027 matched placebo up to the MTD. A total of 2 participants per cohort will be randomized to E2027 matched placebo.
  Interventions: Drug: E2027 matched placebo

INTERVENTIONS:
Drug: E2027 — Participants will receive E2027 capsules, orally once daily (QD) on Days 1 to 14 after an overnight fast of at least 10 hours. E2027 will be administered orally with 240 milliliter (mL) (8 fluid ounces) of water.
  Arms: E2027
Drug: E2027 matched placebo — Participants will receive E2027 matched placebo capsules, orally once daily (QD) on Days 1 to 14 after an overnight fast of at least 10 hours. E2027 matched placebo will be administered orally with 240 mL (8 fluid ounces) of water.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacodynamics (PD) and pharmacokinetics (PK) of multiple ascending oral doses of E2027 in healthy participants.

ELIGIBILITY:
Inclusion Criteria Parts A, B,C and D

1. Nonsmoking, male or female, age ≥50 years and ≤85 years old at the time of informed consent 2. Body mass index (BMI) ≥18 and ≤32 kilogram per square meter (kg/m2) at Screening Part B 3. Born in Japan to Japanese parents and grandparents of Japanese descent 4. Lifestyle, including diet, has not changed significantly since leaving Japan Exclusion Criteria

1. Clinically significant illness that requires medical treatment within 8 weeks or a clinically significant infection that requires medical treatment within 4 weeks of dosing
2. Females who are breastfeeding or pregnant at Screening or Baseline (documented by a negative beta-human chorionic gonadotropin [beta (ß)-hCG] (or human chorionic gonadotropin [hCG]) test with a minimum sensitivity of 25 International Unit per Liter (IU/L) or equivalent units of ß-hCG [or hCG]). A negative urine pregnancy test is required before the administration of the 1st dose per cohort.
3. Females of childbearing potential who:

   * Had unprotected sexual intercourse within 30 days before study entry and do not agree to use a highly effective method of contraception (eg, total abstinence, an intrauterine device, a double barrier method [such as condom plus diaphragm with spermicide] or have a vasectomized partner with confirmed azoospermia but hormonal contraceptives are not permitted) throughout the entire study period and for 28 days after study drug discontinuation
   * Are currently abstinent, and do not agree to use a double barrier method (as described above) or refrain from sexual activity during the study period or for 28 days after study drug discontinuation NOTE: All females will be considered to be of childbearing potential unless they are postmenopausal (amenorrheic for at least 12 consecutive months, in the appropriate age group, and without other known or suspected cause) or have been sterilized surgically (ie, bilateral tubal ligation, total hysterectomy, or bilateral oophorectomy, all with surgery at least 1 month before dosing).
4. Males who have not had a successful vasectomy (confirmed azoospermia) or they and their female partners do not meet the criteria above (ie, not of childbearing potential or practicing highly effective contraception throughout the study period or for 28 days after study drug discontinuation). No sperm donation is allowed during the study period or for 28 days after study drug discontinuation
5. Medical conditions which are not adequately and stably controlled on stable doses of medications or which, in the clinical opinion of the Principal Investigator (PI), may interfere with study procedures or participant safety within 4 weeks before dosing (eg, psychiatric disorders and disorders of the gastrointestinal tract, liver, kidney, respiratory system, endocrine system, hematological system, neurological system, or cardiovascular system, or participants who have a congenital abnormality in metabolism). Participants with the following stable medical conditions, adequately controlled with stable doses of concomitant medications, need not be excluded if in the opinion of the PI, their conditions do not compromise participant safety or study procedures:

   * hypertension without cerebrovascular or cardiovascular complications, controlled on not more than 1 antihypertensive drug
   * hyperlipidemia without cerebrovascular or cardiovascular complications, controlled with diet or monotherapy medication
   * mild, localized diseases of the skin, respiratory tract which do not require systemic medication treatment and without systemic complications
   * mild, localized diseases of the eyes which are not symptomatic and do not require systemic medication treatment and without systemic complications
   * osteoarthritis which does not require opioids for treatment of pain
6. History of cerebrovascular disease (including transient ischemic attack or stroke)
7. Any history of abdominal surgery that may affect pharmacokinetic (PK) profiles of E2027 (eg, hepatectomy, nephrectomy, digestive organ resection) at Screening or Baseline
8. Any other clinically abnormal symptom or organ impairment found by medical history, physical examinations, vital signs, electrocardiogram (ECG) finding, or laboratory test results that requires medical treatment at Screening or Baseline
9. A prolonged QT/QTc interval (QTc >450 millisecond [ms]) demonstrated on ECG at Screening or Baseline (based on average of triplicate ECGs). A history of risk factors for torsade de pointes (eg, heart failure, hypokalemia, family history of long QT Syndrome) or the use of concomitant medications that prolonged the QT/QTc interval
10. Left bundle branch block at Screening or Baseline
11. Persistent systolic blood pressure (BP) >160 millimeter of mercury (mm Hg) or diastolic BP >100 mm Hg at Screening or Baseline (based on BP measured on at least 3 occasions over 2 weeks)
12. Persistent heart rate (HR) less than 50 beats/minute (min) or more than 90 beats/min at Screening or Baseline (based on HR measured on at least 3 occasions over 2 weeks)
13. History of myocardial infarction, ischemic heart disease or cardiac failure
14. History of clinically significant arrhythmia or uncontrolled arrhythmia
15. Known history of clinically significant drug allergy at Screening or Baseline
16. Known history of food allergies or presently experiencing significant seasonal or perennial allergy at Screening or Baseline
17. Known to be human immunodeficiency virus (HIV) positive at Screening
18. Active viral hepatitis (A, B, or C) as demonstrated by positive serology at Screening
19. History of drug or alcohol dependency or abuse within the 2 years before Screening, or those who have a positive urine drug or alcohol test at Screening or Baseline (participants whose positive urine drug test is considered by the investigator and sponsor medical monitor to be due to permitted concomitant medications need not be excluded)
20. Participants who smoke or have used tobacco or nicotine-containing products within 4 weeks before to dosing
21. A Columbia Suicide Severity Rating Scale (C-SSRS) suicidal ideation score of 4 or 5 at Screening or Baseline or for the period within 6 months before to Screening or Baseline or any lifetime suicidal behavior
22. Currently enrolled in another clinical study or used any investigational drug or device within 30 days (or 5 half-lives, whichever is longer) preceding informed consent
23. Engagement in strenuous exercise within 2 weeks before check-in (eg, marathon runners, weight lifters)
24. Any contraindications to cerebrospinal fluid (CSF) sampling by lumbar puncture (LP)
25. Participants with platelet count <60,000, international normalized ratio (INR) >1.2, or partial thromboplastin time (PTT) > upper limit of normal (ULN) at Screening
26. Intake of caffeinated beverages or caffeinated food within 72 hours before dosing
27. Intake of nutritional supplements, juice, and herbal preparations or other foods or beverages that may affect the various drug metabolizing enzymes and transporters (eg, alcohol, grapefruit, grapefruit juice, grapefruit-containing beverages, apple or orange juice, vegetables from the mustard green family [eg, kale, broccoli, watercress, collard greens, kohlrabi, brussel sprouts, mustard], and charbroiled meats) within 1 week before dosing
28. Intake of herbal preparations containing St. John's Wort within 4 weeks before dosing.
29. Intake of over-the-counter (OTC) medications within 14 days (or 5 half-lives, whichever is longer) before dosing unless the principal investigator and sponsor medical monitor consider that they do not compromise participant safety or study assessments
30. Participants who are taking prohibited medications as listed in Concomitant Drug/Therapy section within 14 days before dosing

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2016-08-10 (Actual); Primary Completion 2017-11-29 (Actual); Study Completion 2017-11-29 (Actual)

PRIMARY OUTCOMES:
Maximum drug concentration (Cmax) | Day 1 and Day 14
  Blood samples will be collected on Day 1 at predose and postdose 0.5 (30 minutes), 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 18 hours; Day 14 (at predose and postdose 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 18 hours); and Day 15 (24 hours postdose from Day 14).
Mean predose drug concentration (Cmin) | Predose on Days 2, 4, 6, 8, 10, 12, 13, and 14
Mean time to reach maximum (peak) drug concentration (tmax) | Day 1 and Day 14
  Blood samples will be collected on Day 1 at predose and postdose 0.5 (30 minutes), 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 18 and 24 hours; Day 14 (at predose and postdose 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 18 hours); and Day 15 (24 hours postdose from Day 14).
Mean area under the concentration-time curve from zero time to 24 hours postdose (AUC(0-24h)) | Day 1 and Day 14
  Blood samples will be collected on Day 1 at predose and postdose 0.5 (30 minutes), 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 18 and 24 hours; Day 14 (at predose and postdose 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 18 hours); and Day 15 (24 hours postdose from Day 14).
Mean area under the concentration-time curve from zero time extrapolated to infinity (AUC(0-inf)) | Day 14
  Blood samples will be collected on Day 14 (at predose and postdose 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 18 hours) and Day 15 (24 hours postdose from Day 14).
Mean terminal elimination half-life (t1/2) | Day 14
  Blood samples will be collected on Day 14 (at predose and postdose 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 18 hours) and Day 15 (24 hours postdose from Day 14).
Average steady state drug concentration (Css,av) | Day 14
  Blood samples will be collected on Day 14 (at predose and postdose 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 18 hours) and Day 15 (24 hours postdose from Day 14).
Mean apparent clearance at steady state (CLss/F) | Day 14
  Blood samples will be collected on Day 14 (at predose and postdose 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 18 hours) and Day 15 (24 hours postdose from Day 14).
Mean apparent volume of distribution at steady state (Vss/F) | Day 14
  Blood samples will be collected on Day 14 (at predose and postdose 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 18 hours) and Day 15 (24 hours postdose from Day 14).
Mean accumulation ratio (Rac) (Day 14: Day 1) for AUC(0-24h), Cmax and Cmin | Day 1 and Day 14
  Day 1 at predose and postdose 0.5 (30 minutes), 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 18 and 24 hours; Day 14 (at predose and postdose 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 18 hours); and Day 15 (24 hours postdose from Day 14)
Mean peak-trough fluctuation ratio (PTF) | Day 14
  Blood samples will be collected on Day 14 (at predose and postdose 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, and 18 hours) and Day 15 (24 hours postdose from Day 14).
Mean ratio of cerebrospinal fluid (CSF) : plasma concentrations | Day -2 (time-matched to the Day 13 lumbar puncture [LP]) and Day 13 (predose)

SECONDARY OUTCOMES:
Percentage change from Baseline in pharmacodynamic measure | Day -2 (baseline with no drug) to Day 13 (on drug)
Change from baseline in Observed Fridericia's Correction Formula (QTcF) | Days -1, 1, and 14

CONTACTS AND LOCATIONS:
Locations (1):
- California Clinical Trials Medical Group, Glendale, California, United States